CLINICAL TRIAL: NCT06094296
Title: A Randomized, Double-blind, Phase 2 Study of BMS-986315 and Nivolumab in Combination With Chemotherapy Versus Nivolumab in Combination With Chemotherapy as First-line Treatment for Participants With Stage IV or Recurrent Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Study of BMS-986315 and Nivolumab in Combination With Chemotherapy in Participants With First-line Stage IV or Recurrent Non-small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA047-1009; 2022-503007-22 (EudraCT Number); U1111-1282-5699 (Other: WHO)
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: NSCLC
Keywords: Pharmacokinetics; BMS-986315; Nivolumab; Platinum doublet chemotherapy; NSCLC; Lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Nivolumab; Pemetrexed; Cisplatin; Carboplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1: BMS-986315 Dose Level (DL) 1 + Nivolumab + Histology-based PDCT (Experimental)
  Interventions: Drug: BMS-986315; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin; Drug: Paclitaxel
- Part 1: BMS-986315 DL 2 + Nivolumab + Histology-based PDCT (Experimental)
  Interventions: Drug: BMS-986315; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin; Drug: Paclitaxel
- Part 2: Nivolumab + Histology-based PDCT (Active Comparator)
  Interventions: Drug: Nivolumab; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin; Drug: Paclitaxel
- Part 2: BMS-986315 DL 2 + Nivolumab + Histology-based PDCT (Experimental)
  Interventions: Drug: BMS-986315; Drug: Nivolumab; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin; Drug: Paclitaxel
- Part 2: BMS-986315 DL 1 + Nivolumab + Histology-based PDCT (Experimental)
  Interventions: Drug: BMS-986315; Drug: Nivolumab; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: BMS-986315 — Specified dose on specified days
  Other Names: Anti-NKG2A
  Arms: Part 1: BMS-986315 DL 2 + Nivolumab + Histology-based PDCT; Part 1: BMS-986315 Dose Level (DL) 1 + Nivolumab + Histology-based PDCT; Part 2: BMS-986315 DL 1 + Nivolumab + Histology-based PDCT; Part 2: BMS-986315 DL 2 + Nivolumab + Histology-based PDCT
Drug: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558
  Arms: Part 2: BMS-986315 DL 1 + Nivolumab + Histology-based PDCT; Part 2: BMS-986315 DL 2 + Nivolumab + Histology-based PDCT; Part 2: Nivolumab + Histology-based PDCT
Drug: Pemetrexed — Specified dose on specified days
Drug: Cisplatin — Specified dose on specified days
Drug: Carboplatin — Specified dose on specified days
Drug: Paclitaxel — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of BMS-986315 plus nivolumab in combination with platinum-based doublet chemotherapy (PDCT) versus nivolumab in combination with PDCT in the first-line treatment of Stage IV or recurrent non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have NSCLC with Stage IV or recurrent disease following multimodal therapy for locally advanced disease.
* Study treatment must be first-line therapy for Stage IV or recurrent disease.
* Participants in all parts of the study must have:
* measurable disease per Response Evaluation Criteria in Solid Tumors version 1.1. (RECIST v1.1)
* an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* a life expectancy of at least 3 months at the time of first dose

Exclusion Criteria:

* Untreated symptomatic central nervous system metastases
* Participants with epidermal growth factor receptor (EGFR)/ALK receptor tyrosine kinase (ALK)/ROS proto-oncogene 1 (ROS1)/neurotrophic tyrosine receptor kinase (NTRK)/MET proto-oncogene (MET)/B-Raf proto-oncogene (BRAF)/RET proto-oncogene (RET) mutations amenable to targeted therapies
* Participants with any known medical condition that, in the investigator's opinion, would increase the risk associated with study participation or study drug administration or interfere with the interpretation of safety results

Note: Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (8):
- United States (5):
  - Local Institution - 0038, Glendale, California
  - Local Institution - 0044, Clermont, Florida
  - Local Institution - 0040, Orange City, Florida
  - Local Institution - 0058, Boise, Idaho
  - Local Institution - 0049, Houston, Texas
- Australia (3):
  - Local Institution - 0013, St Leonards, New South Wales
  - Local Institution - 0021, Tweed Heads, New South Wales
  - Local Institution - 0032, Joondalup, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/home

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In Part 1 one participant received study treatment. In Part 2 no participants were enrolled.
Groups:
- Part 1: BMS-986315 + Nivolumab + Histology-based Chemotherapy; Part 2 Arm C: BMS-986315 + Nivolumab + Histology-based Chemotherapy: Participant received BMS-986315 450 mg every 3 weeks in combination with nivolumab 360 mg every 3 weeks plus chemotherapy every 3 weeks
- Part 2 Arm A: Nivolumab + Histology-based Chemotherapy: Participant received Nivolumab 360 mg every 3 weeks plus chemotherapy every 3 weeks
- Part 2 Arm B: BMS-986315 + Nivolumab + Histology-based Chemotherapy: Participant received BMS-986315 900 mg every 3 weeks in combination with nivolumab 360 mg every 3 weeks plus chemotherapy every 3 weeks
Period: Overall Study
Arm/Group | Part 1: BMS-986315 + Nivolumab + Histology-based Chemotherapy | Part 2 Arm A: Nivolumab + Histology-based Chemotherapy | Part 2 Arm B: BMS-986315 + Nivolumab + Histology-based Chemotherapy | Part 2 Arm C: BMS-986315 + Nivolumab + Histology-based Chemotherapy
Started | 1 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Progressive Disease | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: In Part 2, no participants were enrolled, so no analysis was conducted
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: BMS-986315 + Nivolumab + Histology-based Chemotherapy | Part 2 Arm A: Nivolumab + Histology-based Chemotherapy | Part 2 Arm B: BMS-986315 + Nivolumab + Histology-based Chemotherapy | Part 2 Arm C: BMS-986315 + Nivolumab + Histology-based Chemotherapy | Total
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  |  | 0
  Between 18 and 65 years | 1 |  |  |  | 1
  >=65 years | 0 |  |  |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Not providing identifying information to protect participant privacy |  |  |  | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Not providing identifying information to protect participant privacy |  |  |  | NA — Total not calculated because data are not available (NA) in one or more arms.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | NA — Not providing identifying information to protect participant privacy |  |  |  | NA — Total not calculated because data are not available (NA) in one or more arms.
  Not Hispanic or Latino | NA — Not providing identifying information to protect participant privacy |  |  |  | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | NA — Not providing identifying information to protect participant privacy |  |  |  | NA — Total not calculated because data are not available (NA) in one or more arms.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | NA — Not providing identifying information to protect participant privacy |  |  |  | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian | NA — Not providing identifying information to protect participant privacy |  |  |  | NA — Total not calculated because data are not available (NA) in one or more arms.
  Native Hawaiian or Other Pacific Islander | NA — Not providing identifying information to protect participant privacy |  |  |  | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African American | NA — Not providing identifying information to protect participant privacy |  |  |  | NA — Total not calculated because data are not available (NA) in one or more arms.
  White | NA — Not providing identifying information to protect participant privacy |  |  |  | NA — Total not calculated because data are not available (NA) in one or more arms.
  More than one race | NA — Not providing identifying information to protect participant privacy |  |  |  | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | NA — Not providing identifying information to protect participant privacy |  |  |  | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) for Part 1
Description: An adverse event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition occurring in a clinical investigation participant after signing of informed consent, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory test result), symptom, or disease temporally associated with the study intervention.
Time Frame: From first dose through 100 days following last dose of study treatment (assessed for approximately 7 months)
Population: All Treated Participants for Part 1. Pre-specified to be reported for Part 1 only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: BMS-986315 + Nivolumab + Histology-based Chemotherapy
Number analyzed (Participants) | 1
Participants | 1

2. Primary Outcome: Number of Participants With Treatment Related Adverse Events (TRAEs) for Part 1
Description: as for outcome 1
Time Frame: From first dose through 100 days following last dose of study treatment (assessed for approximately 7 months)
Population: All Treated Participants for Part 1. Pre-specified to be reported for Part 1 only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: BMS-986315 + Nivolumab + Histology-based Chemotherapy
Number analyzed (Participants) | 1
Participants | 1

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) for Part 1
Description: Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, and requires inpatient hospitalization or causes prolongation of existing hospitalization.
Time Frame: From first dose through 100 days following last dose of study treatment (assessed for approximately 7 months)
Population: All Treated Participants for Part 1. Pre-specified to be reported for Part 1 only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: BMS-986315 + Nivolumab + Histology-based Chemotherapy
Number analyzed (Participants) | 1
Participants | 0

4. Primary Outcome: Number of Participants With Adverse Events (AEs) Meeting Protocol-defined Dose-limiting Toxicity (DLT) Criteria for Part 1
Description: Dose-Limiting Toxicities (DLTs) are treatment effects serious enough to prevent dose increase.
  Severity grades: 1=Mild, 2=Moderate, 3=Severe, 4=Life-threatening, 5=Death
  * Grade 2 uveitis or eye pain not improving or require systemic treatment
  * Grade 2 pneumonitis or interstitial lung disease >14 days
  * Grade ≥ 3 uveitis, episcleritis, iritis, pneumonitis, bronchospasm or neurologic toxicity
  * Grade 3 colitis not responding >48 hours
  * Hepatic abnormalities without liver metastases: serum transaminases (AST/ALT) >5x & ≤ 8xULN for >2weeks, AST/ALT >8xULN regardless of duration, total bilirubin >3xULN, or concurrent AST/ALT >3xULN & total bilirubin >2xULN
  * Hepatic abnormalities with liver metastases: AST/ALT >8x & ≤10xULN for >2 weeks, AST/ALT >10xULN regardless of duration, total bilirubin > 3xULN, or concurrent AST/ALT >8xULN & total bilirubin >2xULN
  * Grade 3 (hypersensitivity reaction not resolving to Grade 1 in 6 hours; fatigue >7 days; nausea, vomiting, or diarrhea >72 hours)
Time Frame: From first dose (Cycle 1 Day 1) up to day 28
Population: All Treated Participants for Part 1. Pre-specified to be reported for Part 1 only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: BMS-986315 + Nivolumab + Histology-based Chemotherapy
Number analyzed (Participants) | 1
Participants | 0

5. Primary Outcome: Number of Participants With Adverse Events (AEs) Leading to Discontinuation for Part 1
Description: as for outcome 1
Time Frame: From first dose through 100 days following last dose of study treatment (assessed for approximately 7 months)
Population: All Treated Participants for Part 1. Pre-specified to be reported for Part 1 only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: BMS-986315 + Nivolumab + Histology-based Chemotherapy
Number analyzed (Participants) | 1
Participants | 0

6. Primary Outcome: Number of Participants Who Died in Part 1
Description: Number of participants who died during the study
Time Frame: From first dose through 100 days following last dose of study treatment (assessed for approximately 7 months)
Population: All Treated Participants for Part 1. Pre-specified to be reported for Part 1 only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: BMS-986315 + Nivolumab + Histology-based Chemotherapy
Number analyzed (Participants) | 1
Participants | 0

7. Primary Outcome: Objective Response Rate (ORR) for Part 2
Description: Objective response rate (ORR) is defined as the number of participants who achieve a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR), based on blinded independent central review (BICR) assessments using Response Evaluation Criteria in Solid Tumors (RECIST 1.1), divided by the number of all randomized participants.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  No participants were enrolled in Part 2 due to the study termination; therefore, no data were collected for this endpoint.
Time Frame: From randomization until the date of first objectively documented progression or start of subsequent therapy whichever occurred first (planned for up to approximately 5 years)
Population: Pre-specified to be reported for Part 2 only. No participants were enrolled in Part 2 due to the study termination; therefore, no data were collected for this endpoint.
Arm/Group | Part 2 Arm A: Nivolumab + Histology-based Chemotherapy | Part 2 Arm B: BMS-986315 + Nivolumab + Histology-based Chemotherapy | Part 2 Arm C: BMS-986315 + Nivolumab + Histology-based Chemotherapy
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Progression Free Survival (PFS) for Part 2
Description: Progression free survival is defined as the time between the date of randomization and the first date of documented progression, per blinded independent central review (BICR) assessments using Response Evaluation Criteria in Solid Tumors (RECIST 1.1), or death due to any cause, whichever occurs first.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm (Note: The appearance of 1or more new lesions is also considered progression).
  No participants were enrolled in Part 2 due to the study's termination; therefore, no data were collected for this endpoint.
Time Frame: From randomization until the date of first objectively documented progression or death due to any cause, whichever occurred first (planned for up to approximately 5 years)
Population: as for outcome 7
Arm/Group | Part 2 Arm A: Nivolumab + Histology-based Chemotherapy | Part 2 Arm B: BMS-986315 + Nivolumab + Histology-based Chemotherapy | Part 2 Arm C: BMS-986315 + Nivolumab + Histology-based Chemotherapy
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Adverse Events (AEs) for Part 2
Description: An adverse event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition occurring in a clinical investigation participant after signing of informed consent, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory test result), symptom, or disease temporally associated with the study intervention.
  No participants were enrolled in Part 2 due to the study's termination; therefore, no data were collected for this endpoint.
Time Frame: Up to 100 days after discontinuation of study treatment
Population: as for outcome 7
Arm/Group | Part 2 Arm A: Nivolumab + Histology-based Chemotherapy | Part 2 Arm B: BMS-986315 + Nivolumab + Histology-based Chemotherapy | Part 2 Arm C: BMS-986315 + Nivolumab + Histology-based Chemotherapy
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Treatment Related Adverse Events (TRAEs) for Part 2
Description: as for outcome 9
Time Frame: Up to 100 days after discontinuation of study treatment
Population: as for outcome 7
Arm/Group | Part 2 Arm A: Nivolumab + Histology-based Chemotherapy | Part 2 Arm B: BMS-986315 + Nivolumab + Histology-based Chemotherapy | Part 2 Arm C: BMS-986315 + Nivolumab + Histology-based Chemotherapy
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) for Part 2
Description: Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, and requires inpatient hospitalization or causes prolongation of existing hospitalization.
  No participants were enrolled in Part 2 due to the study's termination; therefore, no data were collected for this endpoint.
Time Frame: Up to 100 days after discontinuation of study treatment
Population: as for outcome 7
Arm/Group | Part 2 Arm A: Nivolumab + Histology-based Chemotherapy | Part 2 Arm B: BMS-986315 + Nivolumab + Histology-based Chemotherapy | Part 2 Arm C: BMS-986315 + Nivolumab + Histology-based Chemotherapy
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Adverse Events (AEs) Meeting Protocol-defined Dose-limiting Toxicity (DLT) Criteria for Part 2
Description: as for outcome 4
Time Frame: Up to 100 days after discontinuation of study treatment
Population: as for outcome 7
Arm/Group | Part 2 Arm A: Nivolumab + Histology-based Chemotherapy | Part 2 Arm B: BMS-986315 + Nivolumab + Histology-based Chemotherapy | Part 2 Arm C: BMS-986315 + Nivolumab + Histology-based Chemotherapy
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Adverse Events (AEs) Leading to Discontinuation for Part 2
Description: as for outcome 9
Time Frame: Up to 100 days after discontinuation of study treatment
Population: as for outcome 7
Arm/Group | Part 2 Arm A: Nivolumab + Histology-based Chemotherapy | Part 2 Arm B: BMS-986315 + Nivolumab + Histology-based Chemotherapy | Part 2 Arm C: BMS-986315 + Nivolumab + Histology-based Chemotherapy
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Number of Participants Who Died in Part 2
Description: Number of participants who died during the study
  No participants were enrolled in Part 2 due to the study's termination; therefore, no data were collected for this endpoint.
Time Frame: Up to 100 days after discontinuation of study treatment
Population: as for outcome 7
Arm/Group | Part 2 Arm A: Nivolumab + Histology-based Chemotherapy | Part 2 Arm B: BMS-986315 + Nivolumab + Histology-based Chemotherapy | Part 2 Arm C: BMS-986315 + Nivolumab + Histology-based Chemotherapy
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Duration of Response (DoR) for Part 2
Description: Duration of response is defined as the time between the date of first documented response (CR or PR) that is subsequently confirmed, to the date of the 1st objectively documented tumor progression as determined by BICR (per RECIST 1.1), or death due to any cause, whichever occurs first.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm (Note: The appearance of 1or more new lesions is also considered progression).
Time Frame: as for outcome 8
Population: as for outcome 7
Arm/Group | Part 2 Arm A: Nivolumab + Histology-based Chemotherapy | Part 2 Arm B: BMS-986315 + Nivolumab + Histology-based Chemotherapy | Part 2 Arm C: BMS-986315 + Nivolumab + Histology-based Chemotherapy
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Time to Objective Response (TTR) for Part 2
Description: Time to response (TTR) assessed by BICR is defined as the time between the date of randomization and the first confirmed documented response (CR or PR) per RECIST 1.1 criteria.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  No participants were enrolled in Part 2 due to the study's termination; therefore, no data were collected for this endpoint.
Time Frame: as for outcome 8
Population: as for outcome 7
Arm/Group | Part 2 Arm A: Nivolumab + Histology-based Chemotherapy | Part 2 Arm B: BMS-986315 + Nivolumab + Histology-based Chemotherapy | Part 2 Arm C: BMS-986315 + Nivolumab + Histology-based Chemotherapy
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Disease Control Rate (DCR) for Part 2
Description: Disease control rate (DCR) is defined as the number of participants who achieve a BOR of confirmed CR, confirmed PR, or stable disease (SD), based on BICR assessments (using RECIST 1.1) divided by the number of all randomized participants.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study.
  No participants were enrolled in Part 2 due to the study's termination; therefore, no data were collected for this endpoint.
Time Frame: as for outcome 8
Population: as for outcome 7
Arm/Group | Part 2 Arm A: Nivolumab + Histology-based Chemotherapy | Part 2 Arm B: BMS-986315 + Nivolumab + Histology-based Chemotherapy | Part 2 Arm C: BMS-986315 + Nivolumab + Histology-based Chemotherapy
Number analyzed (Participants) | 0 | 0 | 0

18. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) for Part 2
Description: Cmax is the maximum observed serum concentration.
  No participants were enrolled in Part 2 due to the study's termination; therefore, no data were collected for this endpoint.
Time Frame: Cycle 1 Day 1, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1 (Each Cycle is of 21 Days)
Population: as for outcome 7
Arm/Group | Part 2 Arm A: Nivolumab + Histology-based Chemotherapy | Part 2 Arm B: BMS-986315 + Nivolumab + Histology-based Chemotherapy | Part 2 Arm C: BMS-986315 + Nivolumab + Histology-based Chemotherapy
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Time of Maximum Observed Concentration (Tmax) for Part 2
Description: Tmax is the time of maximum observed serum concentration.
  No participants were enrolled in Part 2 due to the study's termination; therefore, no data were collected for this endpoint.
Time Frame: C1D1, C1D2, C1D4, C1D8, C1D15, C2D1, C3D1, C4D1, C5D1, C5D2, C5D4, C5D8, C5D15, Day 1 of every 4 cycles from cycle 6 (up to 2 years); at 30 and 100 days post last dose (Each Cycle is of 21 Days)
Population: as for outcome 7
Arm/Group | Part 2 Arm A: Nivolumab + Histology-based Chemotherapy | Part 2 Arm B: BMS-986315 + Nivolumab + Histology-based Chemotherapy | Part 2 Arm C: BMS-986315 + Nivolumab + Histology-based Chemotherapy
Number analyzed (Participants) | 0 | 0 | 0

20. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration [AUC(0-T)] for Part 2
Description: AUC (0-T) is the area under the serum concentration-time curve from time zero to time of last quantifiable concentration.
  No participants were enrolled in Part 2 due to the study's termination; therefore, no data were collected for this endpoint.
Time Frame: as for outcome 19
Population: as for outcome 7
Arm/Group | Part 2 Arm A: Nivolumab + Histology-based Chemotherapy | Part 2 Arm B: BMS-986315 + Nivolumab + Histology-based Chemotherapy | Part 2 Arm C: BMS-986315 + Nivolumab + Histology-based Chemotherapy
Number analyzed (Participants) | 0 | 0 | 0

21. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) to BMS-986315 for Part 2
Description: Number of Participants with Anti-drug Antibodies (ADA) to BMS-986315
  No participants were enrolled in Part 2 due to the study's termination; therefore, no data were collected for this endpoint.
Time Frame: Cycle 1 Day 1, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Day 1 of every 4 cycles from cycle 6 (up to 2 years); at 30 and 100 days post last dose (Each Cycle is of 21 Days)
Population: as for outcome 7
Arm/Group | Part 2 Arm A: Nivolumab + Histology-based Chemotherapy | Part 2 Arm B: BMS-986315 + Nivolumab + Histology-based Chemotherapy | Part 2 Arm C: BMS-986315 + Nivolumab + Histology-based Chemotherapy
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-Cause Mortality from first dose until study completion (up to approximately 7 months). SAEs and Other AEs were assessed from first dose through 100 days following last dose of study treatment (up to approximately 7 months).
Description: All-Cause Mortality, Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
  In Part 1 one participant received study treatment. In Part 2 no participants were enrolled.
Arm/Group | Part 1: BMS-986315 + Nivolumab + Histology-based Chemotherapy
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: BMS-986315 + Nivolumab + Histology-based Chemotherapy (N=1)
Anaemia (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/96/NCT06094296/Prot_SAP_000.pdf